CLINICAL TRIAL: NCT00589927
Title: Comparison of Triple Versus Dual Antiplatelet Therapy After ABT578-Eluting Stent Implantation For Long Coronary Lesions
Brief Title: Triple Versus Dual Antiplatelet Therapy After ABT578-Eluting Stent
Acronym: DECLARELONG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CardioVascular Research Foundation, Korea (Other)
Collaborators: Otsuka Korea (Unknown)
Responsible Party: Seong-Wook Park, MD, PhD, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-0003
Record Dates: First submitted 2007-12-31; First posted 2008-01-10 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2009-07

CONDITIONS: Coronary Artery Disease
Keywords: stents; cilostazol
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cilostazol (Experimental): Cilostazol 200mg loading dose within 1 hours after successful stenting, followed by 100mg bid for 8 months
  Interventions: Drug: cilostazol
- placebo (Placebo Comparator): Control placebo 200mg loading dose within 1 hours after successful stenting, followed by 100mg bid for 8 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cilostazol — cilostazol 200mg loading dose within 1 hours after successful stenting, followed by 100mg bid for 8 months
  Arms: cilostazol
Drug: placebo — placebo 200mg loading dose within 1 hours after successful stenting, followed by 100mg bid for 8 months
  Arms: placebo

SUMMARY:
To evaluate whether the cilostazol reduce neointimal hyperplasia after ZES (Zotarolimus-eluting stents) implantation, the investigators performed double-blind,randomized, multicenter, prospective study compared triple antiplatelet therapy (aspirin plus clopidogrel plus cilostazol) and dual antiplatelet therapy (aspirin plus clopidogrel) for 8 months in patients with long coronary lesion treated with ZES.

DETAILED DESCRIPTION:
Use of drug-eluting stent (DES) has reduced the incidence of restenosis rate and the need for repeat revascularization compared to using bare metal stents. DES implantation also significantly reduced the angiographic restenosis in patients with long coronary lesions.However, although the use of DES has decreased the effect of lesion length on restenosis, the restenosis after DES implantation of long coronary lesions remain at a higher risk of restenosis.

Cilostazol, a phosphodiesterase III inhibitor, has been known to reduce smooth muscle proliferation and intimal hyperplasia after endothelial injury and restenosis after balloon angioplasty and bare-metal stent (BMS) implantation when compared with aspirin and clopidogrel or ticlopidine. Recently, the impact of 6-month cilostazol treatment in addition to aspirin and clopidogrel on neointimal hyperplasia after sirolimus-(SES) or paclitaxel-eluting stent (PES) implantation for long-coronary lesions has been evaluated in our institution. It reported that cilostazol treatment achieved primary end point (in-stent late loss) and reduced need of target lesion revascularization without significant adverse drug-side effects with open-label design, which suggest that 6-month treatment of cilostazol effectively inhibits the neointimal hyperplasia after DES implantation and can be safely applied to the patients or lesions with higher risk of restenosis such as diabetes and long lesions.However, our study was done in unblinded manner and might underestimate the angiographic results due to relatively short-term follow-up angiographic follow-up(6-month.

Recently commercially available new-DES, zotarolimus-eluting stent (ZES) demonstrated significant reduction of restenosis and cardiac events during 9-month. However, it has not been tested that 8-month treatment of cilostazol also effectively inhibits the neointimal hyperplasia after ZES implantation in patients with long coronary lesions. Therefore, to evaluate whether the cilostazol reduce neointimal hyperplasia after ZES implantation, the investigators performed double-blind, randomized, multicenter, prospective study compared triple antiplatelet therapy (aspirin plus clopidogrel plus cilostazol) and dual antiplatelet therapy (aspirin plus clopidogrel) for 8 months in patients with long coronary lesion treated with ZES.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical 1) Patients with angina and documented ischemia or patients with documented silent ischemia 2) Patients who are eligible for intracoronary stenting 3) Age >18 years, <75 ages
2. Angiographic 1) De novo lesion 2) Percent diameter stenosis ≥50% 3) Reference vessel size >2.5 mm by visual estimation 4) Lesion length >25 mm by visual estimation that is required for long Endeavor stent implantation (planned total stent length >30mm)

Exclusion Criteria:

1. History of bleeding diathesis or coagulopathy
2. Pregnant
3. Known hypersensitivity or contra-indication to contrast agent, heparin, sirolimus and paclitaxel
4. Limited life-expectancy (less than 1 year) due to combined serious disease
5. ST-elevation acute myocardial infarction
6. Characteristics of lesion 1) Left main disease 2) In-stent restenosis 3) Graft vessels
7. Hematological disease (Neutropenia <3000/mm3, Thrombocytopenia <100,000/mm3)
8. Hepatic dysfunction, liver enzyme (ALT and AST) elevation >3 times normal
9. Renal dysfunction, creatinine >2.0mg/dL
10. Contraindication to aspirin, clopidogrel or cilostazol
11. planned bifurcation stenting

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Angiographic in-stent late loss | 8-months after randomization

SECONDARY OUTCOMES:
Composite of death, MI, and target lesion or vessel revascularization at 12 months, In-stent and in-stent restenosis at 8 months, In-segment late loss at 8 months Adverse side effects during treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Wook Park, MD,PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (10):
- South Korea (10):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Soonchunhyang University Hospital, Cheonan, Cheonan
  - Kangwon National University Hospital, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Hallym University Sacred Heart Hospital,, Pyeongchon
  - Asan Medical Center, Seoul
  - Hangang Sacred Heart Hospital, Seoul
  - Seoul Veterans Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Lee SW, Park SW, Kim YH, Yun SC, Park DW, Lee CW, Kang SJ, Park SJ, Lee JH, Choi SW, Seong IW, Lee NH, Cho YH, Shin WY, Lee SJ, Lee SW, Hyon MS, Bang DW, Choi YJ, Kim HS, Lee BK, Lee K, Park HK, Park CB, Lee SG, Kim MK, Park KH, Park WJ; DECLARE-LONG II Study Investigators. A randomized, double-blind, multicenter comparison study of triple antiplatelet therapy with dual antiplatelet therapy to reduce restenosis after drug-eluting stent implantation in long coronary lesions: results from the DECLARE-LONG II (Drug-Eluting Stenting Followed by Cilostazol Treatment Reduces Late Restenosis in Patients with Long Coronary Lesions) trial. J Am Coll Cardiol. 2011 Mar 15;57(11):1264-70. doi: 10.1016/j.jacc.2010.10.035. PMID 21392640